CLINICAL TRIAL: NCT03878056
Title: Cost-effectiveness Analysis and Patient Safety After Apical Prolapse Surgery by Mesh Via Different Approaches; Vaginal or Robotic-assisted: Multicenter, Prospective Parallel Cohort Study
Brief Title: Cost-effectiveness Comparison Between Vaginal Versus Robotic Mesh Surgery for Apical Prolapse: Prospective, Cohort Study
Acronym: KIDS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Edward Morcos, Principle investigator, Head of Urogynecology, Karolinska Institutet
Other Study IDs: Dnr: 2017/1988-31, 2018/380-32
Record Dates: First submitted 2019-02-14; First posted 2019-03-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Prolapse; Female
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Transvaginal mesh: Vaginal surgery (UpholdTM Lite Vaginal Support, Boston Scientific)
  Interventions: Device: Vaginal: UpholdTM Lite Vaginal Support - Boston Scientific
- Robotic sacral colpopexy: Robotic surgery (Artisyn® Y-Shaped Mesh - Ethicon)
  Interventions: Device: Vaginal: UpholdTM Lite Vaginal Support - Boston Scientific

INTERVENTIONS:
Device: Vaginal: UpholdTM Lite Vaginal Support - Boston Scientific — Apical prolapse reconstructive surgery by Transvaginal mesh vs Robotic sacral colpopexy
  Other Names: Robotic: Artisyn® Y-Shaped Mesh - Ethicon

SUMMARY:
Cost-effectiveness, safety, outcomes and diagnostic development in advanced apical female genital prolapse reconstructive surgery by vaginal and robotic-assisted mesh surgery.

A multicenter, prospective, parallel, cohort, comparative study between the vaginal and robotic-assisted mesh surgery including 200 patients.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common condition and may be disabling and limiting quality of life (QoL) among aging women. POP may arise in the anterior (cystocele), posterior (rectocele) and middle compartment (apical POP) of the vagina. Apical POP includes descent of uterus or vaginal vault (if uterus was previously removed). The lifetime risk of undergoing a single operation for POP or urinary incontinence by age 80 is 11%. In Sweden, the risk to undergo 2 pelvic floor surgery is about 130 000 women. Traditional Surgical repairs of POP using native connective tissues are commonly used but the risk for POP recurrence is high if apical prolapse is present (ca 60%). Thus, minimal invasive surgical approaches by apical trans-vaginal mesh (A-TVM) and robotic sacral colpopexy (RSC) to support the vaginal apex (middle compartment) are in progress. 1 Evidence show effectivity and improved QoL after surgery.

Vaginal and robotic accesses may be available to many patients. Vaginal approach may allow surgeon to perform surgery for all POP compartments and perineal injury in one single surgery opportunity. Contra-indications for general anesthesia and some abdominal diseases or conditions may dismiss the robotic surgery. In contrast, all patients can be operated via the vaginal approach except for patient unwellness. Thus, a direct low cost of vaginal surgery may be possible. In the other hand, costs for robotic surgery are high. Whether or not this may be reflected on cost-effectiveness based on QoL improvement after surgery has not yet been studied.

Visualising synthetic implants i.e. POP mesh and the Tension-Free Vaginal Tape (TVT) implant for urinary incontinence (UI) by ultrasonography (US) has been a subject for some studies. Using US, localisation of the TVT in correlation to urinary bladder neck and how close to urethra may explain outcomes after TVT surgery. Given its importance, knowledge of how mesh anatomical position may influence outcomes, it may be useful in further POP surgery development. Our results indicate that US can be used and is reproducible in mapping of A-TVM (manuscript).

Growing need worldwide is to have more cost-effective and safe health care. Cost-effectiveness, safety, outcomes, POP-recurrence and effects on pelvic floor dysfunction have not yet been directly compared between vaginal and robotic mesh surgery for apical POP.

Topic: Cost-Effectiveness (Vaginal vs robotic POP mesh surgery), QoL, safety and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Posthysterectomy prolapse of the vaginal apex, with or without cystocele/rectocele, where the vaginal apex descends at least 50% of the total vaginal length
* Uterine prolapse, with or without cystocele/rectocele, where the leading edge of the cervix descends at least 50% of the total vaginal length and TVL minus point C= ≤ 2 cm
* Prolapse specific pelvic symptom of pelvic heaviness and/or vaginal bulging
* Reproductive years in the past (biologically or reproductive decision)
* Being able to make an informed consent on participation
* Physically and cognitively capable of participating in the required follow-up
* No exclusion criteria fulfilled

Exclusion Criteria:

* Posthysterectomy prolapse of the vaginal apex where the vaginal apex descends less than 50% of the total vaginal length regardless of whether a cystocele/rectocele is present or not
* Uterine prolapse, with or without cystocele, where the leading edge of the cervix descends less than 50% of the total vaginal length
* If cervix elongation is present corresponding to: TVL minus point C= >2 cm without uterine prolapse.
* If prolapse specific pelvic symptoms of pelvic heaviness and/or vaginal bulging are not present
* Previous or current pelvic organ cancer (regardless of treatment)
* Severe rheumatic disease
* Insulin treated severe diabetes mellitus
* Connective tissue disorders (SLE, Sjögrens syndrome, Marfans syndrome, Ehlers Danlos, collagenosis, polymyositis or rheumatic myalgia)
* Current systemic steroid treatment
* Other clinically relevant pelvic disorders for which surgery is indicated including stress urinary incontinence.
* Decision to perform prolapse surgery using other medical devices/mesh

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women (female)
Study Population: Women with apical prolapse and suffering prolapse symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness measurements and comparison between vaginal and robotic mesh surgery for apical prolapse | Changes from baseline an up to 1, 5 and 10 years
  Cost-effectiveness analysis: cost-effectiveness will be evaluated by comparing the vaginal approach with the robotic approach in term of incremental costs and incremental benefits (measured by QALYs gained).15 The incremental cost-effectiveness ratio (ICER) gives the marginal cost for each additional QALY gained by treating a patient using the robotic approach compared to the vaginal approach. To evaluate cost-effectiveness, the ICER must be compared with a reference willingness to pay (WTP) value. Sweden has no such official number, but the National Institute of Clinical Excellence (NICE) in the United Kingdom states a willingness to pay between 20,000 - 30,000 British pounds. If the ICER is below this threshold, the robotic approach will be considered cost-effective compared to the vaginal approach.

SECONDARY OUTCOMES:
Measurement of anatomical outcomes by Pelvic Organ Prolapse Quantification system (POP-Q): vaginal mesh utero-/colpopexy vs Robotic Sacral Colpopexy | Changes from baseline an up to 3 months, 1, 5 and 10 years
  Grading of genital prolapse will be performed using the pelvic organ prolapse quantification (POP-Q) system which is a quantitative method for the assessment of vaginal topography and conforms to the standards recommended by the International Continence Society as described by Bump et al. (Am J Obstetrics Gynecology1996). Postoperative examinations are to be performed by the trial gynecologist with the patient in a supine position. Prolapse of the middle compartment equivalent to, or more, than 50% of the total vaginal length (TVL) (i.e. point C positioned at, or distal to, a point between the hymen and half the total vaginal length) is required for inclusion of a patient in the trial.
Measurement of generic quality of Life (QoL) by The 15D instrument of health-related quality of Life (15D): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  The 15D is a generic, comprehensive, self-administered, 15-dimensional, preference-based questionnaire. The 15D includes 15-dimensions: mobility, vision, hearing, breathing, sleeping, eating, speech (communication), excretion, usual activity, mental function, discomfort, depression, distress, vitality, and sexual functions. Each dimension has five descriptive levels to choose from. The 15D can be used as a profile and a single index score measure. The valuation system is based on the application of multi-attribute utility theory. The single index or utility score represents the generic health-related quality of life on a maximum value of 1 (full health) to lower bound of 0 (being dead). From the 15D, the generic minimal important change (MIC) can be calculated to indicate improvement or deterioration. Also, he quality adjusted life-year (QALY) is evaluated using the estimated 15D values preoperative and after surgery.
Measurement of pelvic floor symptoms by Pelvic Floor Distress Inventory (PFDI-20): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  The PFDI-20 is both a symptom inventory and a measure of the degree of bother and distress (quality-of-life) caused by pelvic floor symptoms. It is a short-form version of the Pelvic Floor Distress Inventory. The questionnaire has been validated for use in pelvic reconstructive surgery and has proven sensitive to change.
  The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions.
Ultrasound measurement of mesh length in cm and mapping of mesh in correlation to bladder and urethra: vaginal mesh utero-/colpopexy vs Robotic Sacral | Ultrasound measurements at 1, 5 and 10 years after surgery
  2D, 3D ultrasound mapping of prolapse mesh length in cm and mesh position from the urinary bladder neck and urethra as measured in cm. Further, to investigate if mesh position correlate to urinary incontinence and/or bladder emptying difficulties (urinary retention).
Measurement of generic QoL by health related quality of life by EuroQol 5-dimensions questionnaire (EQ-5D): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  The EQ-5D questionnaire is used to assess the health condition. It is an instrument to be used to measure generic quality of life in a similar way to 15D, and will be used to measure adjusted quality of life (QALYs). Similar to the 15D, the questionnaire results are mapped to a single utility value.
Measurement of life impact in women with pelvic floor disorders by Pelvic Floor Impact Questionnaire-short form 7 (PFIQ-7): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  The PFIQ-7 is an abridged version of the PFIQ and is used to assess life impact in women with pelvic floor disorders. The PFIQ-7 summary score is calculated by adding the scores from the 3 scales together to obtain the summary score (range 0-300).
Measurement of sexual function by Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  The validated PISQ-12 is a condition-specific, 12-item questionnaire on sexual function, with ordinal response alternatives based on a 5-point Likert scale. The PISQ-12 correlates well with other sexual health questionnaires and has shown sensitivity to change after pelvic reconstructive surgery and predictability of scores using the unabridged PISQ (31 items). The specific questions can be combined to form a score where higher scores indicate better sexual function. The maximum PISQ-12 score is 48. The twelve questions of the PISQ-12 can be divided into three domains: behavioral-emotive, partner-related and physical.
Measurement of Pain by patient self-reporting Visual analogue scale (VAS-scale): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of pain.
Measurement of urinary incontinence by patient self-reporting Visual analogue scale (VAS-scale): vaginal mesh utero-/colpopexy vs Robotic Sacral | Changes from baseline an up to15 days, 3,6&9 months, 1-5 and 10 years
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of severity of urinary incontinence. VAS scale for urinary incontinence: 0 indicate no urinary incontinence whereas 10 indicates maximal or severe urinary incontinence.
Measurement of patient satisfaction by patient self-reporting Visual analogue scale (VAS-scale): vaginal mesh utero-/colpopexy vs Robotic Sacral | Assessment after operation: 15 days, 3,6&9 months, 1-5 and 10 years
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of satisfaction after mesh surgery. VAS scale for patient satisfaction: 0 indicates no satisfaction whereas 10 indicates maximal satisfaction.
Measurement of patient recommendation to other patients to undergo same surgery if they suffer apical prolapse (assessed by patient self-reporting Visual analogue scale (VAS-scale): vaginal mesh utero-/colpopexy vs Robotic Sacral | Assessment after operation: 15 days, 3,6&9 months, 1-5 and 10 years
  VAS scale is a numeric rating scale and ranges from 0-10 (each digit is 1cm) where 0 indicates no and 10 indicates maximum, digits between 0-10 indicate degree of satisfaction. VAS scale for patient recommendation to other patients to undergo same surgery if they suffer apical prolapse: 0 indicates no recommendation whereas 10 indicates maximal recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Morcos, MD, PhD, Principal Investigator — Karolinska Institutet Danderyds Sjukhus (KIDS)
Locations (1):
- Division of Obstetrics and Gynecology, Department of Clinical Sciences, Karolinska Institutet Danderyd University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided